CLINICAL TRIAL: NCT02851667
Title: Promoting Family Health, Happiness, and Harmony Through a Community-based "Learning Family" Campaign
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Lam Tai-Hing, Chair Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UW10-415
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Training group (Experimental): Resident training programs such as talks, day camp and thematic activities were delivered in training group.
  Interventions: Behavioral: Resident training programs

INTERVENTIONS:
Behavioral: Resident training programs — A total of 24 resident training programs such as talks, day camp and thematic activities were delivered in the intervention estate by CFSC from June to November 2011. Each program included an introduction to the concepts of Learning Family and family 3Hs as well as how to promote family 3Hs through learning and communicating with family, delivered by interactive games and workshops.

SUMMARY:
According to the Social Welfare Department statistics, Kwun Tong has been ranked as the highest for the reported cases of elderly abuse (12.3%), the second and fourth highest for the reported cases of battered spouse (9.2%) and child abuse (7.9%) respectively. To strengthen family well-being in the Kwun Tong community, the investigators adopt a community-based participatory (CBP) approach and implement a community-based "Learning Family" campaign in Kwun Tong district with the investigators collaborator, the Christian Family Service Centre (CFSC). The campaign aims to promote family health, happiness, and harmony (3Hs) through cultivating cooperative and self-regulated family learning culture in Kwun Tong district.

DETAILED DESCRIPTION:
Family well-being, which has been conceptualized as "family-life satisfaction", "sense of well-being" and "family function", is associated with outcomes such as hypertension, self-rated health, depression, and self-esteem in family members. Interpersonal harmony in the family is believed to be crucial for the Chinese who see it as contributing not only to each individual member's welfare but also to a well-organized and peaceful world. According to traditional Confucius ideals, family harmony is the basis for an individual's happiness. The investigators qualitative studies in Hong Kong have also found that family health, happiness and harmony (3Hs) are three major themes of family well-being. Family health includes physical and mental health of family members, which is strongly related to psychological capital and family unity. Family happiness can be enhanced by spending time with family members and building connection with friends and relatives. Family harmony means absence of conflicts and effective communication with family members. Forbearance and spending time with family are important in forming a harmonious family.

Learning Families Project was initiated based on the social ecological model. Social ecological model is a framework to examine the dynamic interrelations among various personal and environmental factors. This model emphasizes people's behaviors are affected by factors of different levels including intra-personal, inter-personal, community and societal factors. These programs promoted the concepts of Learning Family and family 3Hs to the participants (intra-personal level). The concepts of Learning Family indicated that family relationship could be improved when family members learnt something together. These programs also provided a platform for family members to learn together and communicate with each other (inter-personal level), as well as for residents to interact in these community activities (community level).

ELIGIBILITY:
Inclusion Criteria:

* Residents living in the intervention estate
* Hong Kong residents
* Older than 10 years of age
* Could communicate in Chinese (Cantonese or Putonghua)

Exclusion Criteria:

* Participants who fail to meet the inclusion criteria

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 980 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Changes in family communication time from baseline to 6 weeks after intervention | Baseline and 6 weeks after intervention
  Family communication time (minutes per day) was assessed.
Changes in perceived communication adequacy from baseline to 6 weeks after intervention | Baseline and 6 weeks after intervention
  Perceived communication adequacy was assessed by a 1-5 score.
Changes in family harmony from baseline to 6 weeks after intervention | Baseline and 6 weeks after intervention
  Family harmony was assessed by a 0-10 score.
Changes in family happiness from baseline to 6 weeks after intervention | Baseline and 6 weeks after intervention
  Family happiness was assessed by a 0-10 score.
Changes in family health from baseline to 6 weeks after intervention | Baseline and 6 weeks after intervention
  Family health was assessed by a 0-10 score.

SECONDARY OUTCOMES:
Changes in neighborhood cohesion from baseline to 1 year after intervention | Baseline and 1 year after intervention
  Neighborhood cohesion was assessed by a 5-items scale.

CONTACTS AND LOCATIONS:
Overall Officials: Tai Hing Lam, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Christian Family Service Center, Hong Kong, Hong Kong

REFERENCES:
- [Background] Berge JM, Mendenhall TJ, Doherty WJ. Using Community-based Participatory Research (CBPR) To Target Health Disparities in Families. Fam Relat. 2009 Oct 1;58(4):475-488. doi: 10.1111/j.1741-3729.2009.00567.x. PMID 20625444
- [Background] Macaulay AC. Promoting participatory research by family physicians. Ann Fam Med. 2007 Nov-Dec;5(6):557-60. doi: 10.1370/afm.755. PMID 18025494
- [Background] White GW, Suchowierska M, Campbell M. Developing and systematically implementing participatory action research. Arch Phys Med Rehabil. 2004 Apr;85(4 Suppl 2):S3-12. doi: 10.1016/j.apmr.2003.08.109. PMID 15083417
- [Background] Lam WW, Fielding R, McDowell I, Johnston J, Chan S, Leung GM, Lam TH. Perspectives on family health, happiness and harmony (3H) among Hong Kong Chinese people: a qualitative study. Health Educ Res. 2012 Oct;27(5):767-79. doi: 10.1093/her/cys087. Epub 2012 Aug 20. PMID 22907531
- [Derived] Shen C, Wan A, Kwok LT, Pang S, Wang X, Stewart SM, Lam TH, Chan SSC. A Community-Based Intervention Program to Enhance Family Communication and Family Well-being: The Learning Families Project in Hong Kong. Front Public Health. 2017 Sep 29;5:257. doi: 10.3389/fpubh.2017.00257. eCollection 2017. PMID 29085815
- [Derived] Shen C, Wan A, Kwok LT, Pang S, Wang X, Stewart SM, Lam TH, Chan SS. A community based intervention program to enhance neighborhood cohesion: The Learning Families Project in Hong Kong. PLoS One. 2017 Aug 21;12(8):e0182722. doi: 10.1371/journal.pone.0182722. eCollection 2017. PMID 28827798